CLINICAL TRIAL: NCT07168239
Title: Effectiveness of Nursing Educational Intervention on Vascular Access Self-Care in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Ana Catarina Silva, Registered Nurse, Aveiro University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Diaverum08072024
Record Dates: First submitted 2025-08-13; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease Patients on Hemodialysis

STUDY DESIGN:
Intervention Model Description: INTERVENTIONAL STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients from two Hemodialysis units with AVF as Vascular Access (Experimental): Population of CKD patients undergoing HD from two portuguese HD units. The sample was non-probabilistic and convenience-based, including patients with an AVF in use. A set of health education sessions were developed for patients who did not exhibit fully adequate behaviour in the first assessment of the Scale of Assessment of Self-Care with AVF in HD.
  Interventions: Behavioral: ENHANCING VASCULAR ACCESS SELF-CARE IN HEMODIALYSIS PATIENTS

INTERVENTIONS:
Behavioral: ENHANCING VASCULAR ACCESS SELF-CARE IN HEMODIALYSIS PATIENTS — A set of health education sessions were developed for patients who did not exhibit fully adequate behaviour in the first assessment of the Scale of Assessment of Self-Care with AVF in HD. The sessions were conducted individually through an expository method and providing an informative leaflet. The sessions focused on the areas presented by the scale, i.e. prevention of thrombosis and infection, signs and symptoms of intra/interdialytic complications, haemostasis care, protection of the AV limb and correct assessment of signs and symptoms suggestive of complications with the AVF, evaluation of AVF functionality and detection of thrombosis, changes in colour and sensitivity of the hand corresponding to the AV, pain in the AV limb

SUMMARY:
Background: Hemodialysis patients experience health-illness transitions, which are prompted by changes in social and personal roles as they adapt to chronic kidney disease and its treatments. In this context, nurses play a facilitative role in supporting these transitions, aiming to enhance the patients' sense of well-being.

There is an increasing need to provide care that positively impacts clinical and health outcomes, including the empowerment of these patients to be as independent as possible including promoting self-care for their vascular access.

The present study aims to assess the self-care profile regarding vascular access in a population of patients with chronic kidney disease undergoing outpatient hemodialysis and to evaluate the impact of educational nursing interventions on the transition process to self-care with vascular access in this population.

Methods: The investigators conducted a prospective, quantitative, and cross-sectional study with an interventional methodology, which involved an initial diagnostic assessment about self-care behaviours with the arteriovenous fistula, followed by an educational intervention to promote adherence to self-care, and a subsequent re-evaluation of the outcomes after the intervention. The assessment of self-care behaviours with the arteriovenous fistula was carried out by the Self-Care Behaviour Assessment Scale with arteriovenous fistula in Hemodialysis.

Data collection was split in three parts: sociodemographic characterization, clinical characterization of participants, and assessment of self-care behaviours with the AVF.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients on outpatient HD
* Independent in self-care
* With AVF as Vascular Access

Exclusion Criteria:

* Usage of CVC or AVP as Vascular Access
* Cognitive impairment (assessed through the Mini-Mental State Examination developed by Folstein et al., 1975)
* non-fluent in Portuguese language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Self-care behaviours with the arteriovenous fistula after a nursing intervention | 3 months
  Data collection of self-care behaviours with the AVF, as described for the primary outcomes, after a nursing intervention.
  Inferential statistical analyses were performed. A paired t-test was used to compare participants' knowledge levels ie. overall score, score on signs and symptoms, and score on complication prevention, at two distinct points.

SECONDARY OUTCOMES:
Self-care behaviours with the AVF | 1 month
  Carried out with the Scale of Assessment of Self-Care with AVF in HD. This scale consists of 16 items, with a two-dimensional structure with a total value of Cronbach's alpha of 0.797. The two subscales are management of signs and symptoms and prevention of complications.
  The scale comprises 31 items scored on a five-point Likert scale, ranging from 31 to 155 points overall. Lower scores reflect insufficient or inconsistent self-care behaviors, while higher scores indicate greater adequacy and consistency in knowledge, attitudes, and practices The application of the scale can be segmented by domain to identify areas with potential for intervention, while the overall score provides an overview of the patient's autonomy in these behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Catarina Brito Silva, Master, Principal Investigator — Student
Locations (1):
- Universidade de Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT07168239/Prot_SAP_ICF_000.pdf